CLINICAL TRIAL: NCT06782581
Title: Positive Activities for Asian American Cancer Patients and Caregivers
Brief Title: CARE Study: Cancer, Asian Americans, and Relationship Enrichment
Acronym: CARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Lilian Shin-Cho, Principal Investigator, Assistant Professor, Fox Chase Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 24-1006; 5R00CA267678-04 (NIH)
Record Dates: First submitted 2024-09-06; First posted 2025-01-20 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Neoplasm
Keywords: Asian American; Cancer; Patient; Positive Activities; Well-being; Caregiver
MeSH Terms: conditions — Neoplasms | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contribution (Experimental): Contribution to caregiver wellbeing via household tasks. If the household contribution condition is chosen, participants will be given instructions and examples/list of things they could do to contribute to the well-being of their caregiver (e.g., cook a meal, take pet for a walk, water the plants). If the outside contribution condition is chosen, participants will be given instructions and examples/list of things they could do to contribute to the world outside of their own home (e.g., pick up litter in neighborhood, buy coffee for stranger, donate food/clothing to homeless)
  Interventions: Behavioral: Contribution to Caregivers Well-Being
- Control Group (Placebo Comparator): Participants in the control group will be asked to factually describe either (1) immediate environment, (2) the weather, or (3) organization of closet
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Contribution to Caregivers Well-Being — Contribute to caregiver's well-being via household tasks.
  Other Names: Household Contribution; Internal Contribution
  Arms: Contribution
Behavioral: Control — factually describe either (1) immediate environment, (2) the weather, or (3) organization of closet
  Other Names: Experimental Arm; Control Group
  Arms: Control Group

SUMMARY:
The overarching goal of the current study is to reduce the burden Asian American patients may feel are on their caregivers by designing and testing the feasibility and efficacy of a positive activity intervention designed to increase a sense of autonomy, competence, and connectedness, each of which have been shown to be associated with psychological benefits according to self-determination theory.

DETAILED DESCRIPTION:
This study will introduce two new positive activities, household contribution and outside contribution, which have been specifically created for AA cancer patients and have not been previously investigated. These interventions have been developed with consideration of culture-related challenges, Hofstede's concept of collectivist cultures, and self-determination theory. This study will be the first randomized controlled trial to assess the impact of these new positive activities on Asian-American cancer patients.

ELIGIBILITY:
Inclusion Criteria for Patients:

1. self-identifies as Asian American or Asian
2. males or females ages 21-80 years
3. within 2 years of any cancer diagnosis or stage 4 cancer diagnosis
4. actively undergoing surgery or systemic therapy (e.g., chemotherapy, radiation, immunotherapy) or within the past 6 months,
5. able to identify a caregiver (e.g., spouse) who lives in the same household or see at least 3 times per week
6. able to read, write, and speak English (i.e., English proficient; EP) or Mandarin/simplified Chinese.

Exclusion Criteria for patients:

1. life expectancy less than 6 months in the opinion of the primary physician
2. inability to stand or walk on their own or other physical limitations that preclude them from participating (3+ on ECOG performance status),
3. major thought disorder (e.g., schizophrenia or bipolar [patient records or self-disclosure]).

Inclusion Criteria for Caregivers:

1. identifies as Asian American or Asian,
2. patient considers them to be caregiver
3. English proficient or Mandarin Chinese proficient
4. access to computer/phone, internet, and web browser.

Exclusion Criteria for Caregivers:

1. unwilling or unable to participate in the study for any reason,
2. under the age of 18.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Affect-Adjective Scale (modified) (AAS) | Baseline/pre-intervention, midpoint/during the intervention (2 weeks), immediately after the intervention (4 weeks), and follow-up 4 weeks after the intervention (8 weeks)
  Primary Outcome Measure: affective well-being
  scores range from 0-6, with 6 indicating higher negative or positive affect
Patient-Reported Outcomes Measurement Information System Global Health (PROMIS G10) | Baseline/pre-intervention, midpoint/during the intervention (2 weeks), immediately after the intervention (4 weeks), and follow-up 4 weeks after the intervention (8 weeks)
  Primary Outcome Measure: health-related quality of life
  scores range from 3 to 15, with higher scores indicating better physical health scores range from 4 to 20, with high scores indicating better mental health

SECONDARY OUTCOMES:
Balanced Measure of Psychological Needs (BMPN) | Baseline/pre-intervention, midpoint/during the intervention (2 weeks), immediately after the intervention (4 weeks), and follow-up 4 weeks after the intervention (8 weeks)
  Secondary Outcome Measure: autonomy, competence, and connectedness
  scores range from 1 to 5, with higher scores indicating more autonomy, competence, or connectedness
Self-Perceived Burden Scale | Baseline/pre-intervention, midpoint/during the intervention (2 weeks), immediately after the intervention (4 weeks), and follow-up 4 weeks after the intervention (8 weeks)
  Secondary Outcome Measure: perceived burdensomeness
  scores range from 10 to 50, with higher scores indicating more self-perceived burdensomeness

OTHER OUTCOMES:
Perceived Stress Scale (PSS) | Baseline/pre-intervention, midpoint/during the intervention (2 weeks), immediately after the intervention (4 weeks), and follow-up 4 weeks after the intervention(8 weeks)
  Other Pre-specified Outcome Measure: patient stres
  PSS: scores range from 0 to 16, with higher scores indicating more stress
PROMIS Patient-Reported Outcomes Measurement Information System Depression 4a (PROMIS Depr4a) | Baseline/pre-intervention, midpoint/during the intervention (2 weeks), immediately after the intervention (4 weeks), and follow-up 4 weeks after the intervention(8 weeks)
  Other Pre-specified Outcome Measure: depression
  PROMIS Depr4a: scores range from 4 to 20 with higher scores indicating more depressive symptoms
MD Anderson Symptom Inventory (MDASI) | Baseline/pre-intervention, midpoint/during the intervention (2 weeks), immediately after the intervention (4 weeks), and follow-up 4 weeks after the intervention(8 weeks)
  Other Pre-specified Outcome Measure: clinical symptoms
  MDASI: scores range from 0 to 10 with higher scores indicating more symptoms or more interference
Getting Along Scale | Baseline/pre-intervention, midpoint/during the intervention (2 weeks), immediately after the intervention (4 weeks), and follow-up 4 weeks after the intervention(8 weeks)
  Other Pre-specified Outcome Measure: interpersonal well-being
  Getting Along: scores range from 4 to 16, with higher scores indicating getting along better

CONTACTS AND LOCATIONS:
Locations (1):
- Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania, United States